CLINICAL TRIAL: NCT04955561
Title: CO2-Patterns During Hyperoxia and Physical Exercise in People With Severe COPD - a Randomized, Double-blind Cross Over Trial
Brief Title: CO2-Patterns During Hyperoxia and Physical Exercise in COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Responsible Party: Principal Investigator, Klaus Kenn, Principal Investigator, Philipps University Marburg
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CO2-Hyperoxia & Exercise
Record Dates: First submitted 2021-05-04; First posted 2021-07-09 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: COPD
Keywords: CO2; oxygen; walking exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Oxygen; Air

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Randomised to begin with oxygen-supplementation at 10L/min during ESWT (Experimental): Randomised order of tests starting with the 10L/min O2, during the ESWT followed by prescribed O2 flow rate or medical air in randomised order on seperate days
  Interventions: Other: Oxygen therapy; Other: Medical Air; Other: 10L/min O2
- Randomised to begin with medical air supplementation at prescibed O2 flow rate during ESWT (Experimental): Randomised order of tests starting with the medical air during the ESWT followed by prescribed O2 flow rate or 10L/min O2 in randomised order on seperate days
  Interventions: Other: Oxygen therapy; Other: Medical Air; Other: 10L/min O2
- Randomised to begin with oxygen supplementation at prescibed O2 flow rate during ESWT (Experimental): Randomised order of tests starting with the prescribed O2 flow rate, during the ESWT followed by 10L/min O2 or medical air in randomised order on seperate days
  Interventions: Other: Oxygen therapy; Other: Medical Air; Other: 10L/min O2

INTERVENTIONS:
Other: Oxygen therapy — Supplemental O2 at rest of 10 l/min for ten minutes followed by supplemental O2 at the prescribed exercise O2-flow rate during ESWT.
Other: Medical Air — Supplemental O2 at rest of 10 l/min for ten minutes followed by medical Air at prescribed O2 flow rate during ESWT.
Other: 10L/min O2 — Supplemental O2 at rest of 10 l/min for ten minutes followed by 10L/min O2 during ESWT.

SUMMARY:
The aim of the study is to investigate a possible correlation between the change in PCO2 during a hyperoxia-test and the change in PCO2 during walking in people with COPD

DETAILED DESCRIPTION:
Rationale:

Carbon dioxide partial pressure (PCO2) varies significantly in patients with advanced chronic obstructive pulmonary disease (COPD). Data from the Swedish LTOT Registry showed that PCO2 is an independent predictor for mortality and that there is a U-shaped relationship. Patients with advanced COPD who are still normocapnic at rest may still develop a clinically relevant, exercise-induced carbon dioxide (CO2) retention during exercise/ activity. It is also known that altered breathing patterns at night in COPD patients can lead to nocturnal hypercapnia, especially during REM sleep. The course of PCO2 cannot be reliably predicted by lung function parameters or resting blood gas analysis. Since exercise tests with blood gas control or nightly PCO2 monitoring are rarely performed in clinical routine, exercise induced CO2 retention often remains undetected. In the literature, there is little information on PCO2 behaviour under everyday conditions (with or without LTOT) such as rest, physical exertion and nightly sleep. Therefore, predictors that could describe the PCO2 patterns are missing. However, one former study by O'Donnel from 2002 showed that the change in CO2 under hyperoxia conditions could provide predictive information for the change in CO2 with exercise.

Objective:

Primary aim of this study is to investigate whether the change of PCO2 during a hyperoxia-test (10l/min O2 at rest) correlates with the change of PCO2 during walking exercise with either a: l/min O2 as prescribed; b: medical air; c: 10l/min O2.

Design:

This study is a randomized, controlled cross-over trial. Following an initial maximal incremental shuttle walk test (ISWT), the participant will perform 3 endurance shuttle walk tests (ESWT) at 85% of the maximum ISWT pace on three consecutive days (24h break between ESWTs). In a randomized order, participants will perform one ESWTs with O2-flow as prescribed (e.g. study day 1), one with medical air (same flow rate as prescribed oxygen) (e.g. study day 2) and one with 10l/min O2 (e.g. study day 3). An additional hyperoxia test (10l/min O2 for ten minutes; at resting condition) will be perfomed on each day prior to performing an ESWT.

ELIGIBILITY:
Inclusion Criteria:

* COPD III/ IV
* 35mmHg < PCO2 <= 55mmHg (under resting conditions, breathing room air)
* Hypoxemia (PaO2<60mmHg) under room air conditions (rest or during exercise) or SpO2 <88% during exercise
* established oxygen therapy or given indication for oxygen therapy
* written informed consent

Exclusion Criteria:

* acute exacerbation of COPD
* exercise limiting cardiac or orthopedic comorbidites
* PaO2 <50mmHg at rest, breathing room air

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-07-13 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Change in PCO2 during hyperoxia at rest | Change from baseline to after 10 minutes breathing 10L/min oxygen
  pCO2 measured by capillary blood gases taken before and after the hyperoxia test
Change in PCO2 from rest to end exercise (endurance shuttle walk test) | Change from baseline to the end of the ESWT, up to 20 minutes
  pCO2 measured by capillary blood gases taken before and after the ESWT

SECONDARY OUTCOMES:
Transcutaneous partial pressure of CO2 (TcPCO2) during hyperoxia test | Continuously from baseline to 10 minutes breathing 10L/min oxygen
  TcPCO2 measured by continuous transcutaneous recording via Sentec-Digital Monitor® (Sentec, Therwil, Switzerland)
Transcutaneous partial pressure of CO2 (TcPCO2) during endurance shuttle walk test | Continuously during ESWT, up to 20 minutes
  TcPCO2 measured by continuous transcutaneous recording via Sentec-Digital Monitor® (Sentec, Therwil, Switzerland)
Breathing frequency during hyperoxia test | Continuously from baseline to 10 minutes breathing 10L/min oxygen
  Breathing frequency during the hyperoxia test measured by ApneaLink Air™ (ResMed)
Breathing frequency during endurance shuttle walk test | Continuously during ESWT, up to 20 minutes
  Breathing frequency during the ESWT measured by ApneaLink Air™ (ResMed)
Heart rate during endurance shuttle walk test | Continuously during ESWT, up to 20 minutes
  Heart rate measured by continuous transcutaneous recordung via Sentec-Digital Monitor® (Sentec, Therwil, Switzerland)
Heart rate during hyperoxia test | Continuously from baseline to 10 minutes breathing 10L/min oxygen
  Heart rate measured by continuous transcutaneous recordung via Sentec-Digital Monitor® (Sentec, Therwil, Switzerland)
Change of capillary partial pressure of O2 (pO2) during endurance shuttle walk test | Change from baseline to the end of the ESWT, up to 20 minutes
  pO2 measured by capillary blood gases taken before and after the ESWT
Change of inspiratory capacity during endurance shuttle walk test | Change from baseline to the end of the ESWT, up to 20 minutes
  IC measured by SpiroSense (Pari) before and after the ESWT

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Berchtesgadener Land, Schön Kliniken, Schönau am Königssee, Germany

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF